CLINICAL TRIAL: NCT03603743
Title: Efficacy of High Intensity Interval Training vs Moderate Intensity and Continuous Training on Autonomic Nervous System Modulations in Chronic Heart Failure
Brief Title: High Intensity Interval Training vs Moderate Intensity and Continuous Training in Chronic Heart Failure
Acronym: HRVFIT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiovascular and Pulmonary Rehabilitation Center of Saint Orens (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University Hospital, Toulouse (Other); Clinique Pasteur (Other)
Responsible Party: Principal Investigator, Lisa RICHARD, MD, Principal Investigator, Cardiologist, Cardiovascular and Pulmonary Rehabilitation Center of Saint Orens
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2-15-12
Record Dates: First submitted 2018-07-13; First posted 2018-07-27 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Chronic Heart Failure
Keywords: exercise training; chronic heart failure; parasympathetic; autonomic nervous system; cardiorespiratory fitness; cardiac rehabilitation
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: subjects were randomly assigned to one of the two groups:
  1. high intensity interval training
  2. moderate intensity and continuous training Block size = 4, allocation ratio 1:1
Who Masked: Investigator, Outcomes Assessor
Masking Description: heart rate variability analyses and echocardiography were performed by investigators blind to randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high intensity interval training (Experimental): high intensity interval training: two sets of 8-min intervals at 100% of peak power output (PPO). Each interval set was composed of repeated bouts of 30 s at 100% of PPO interspersed by 30 s of passive recovery in the seated position. Four minutes of passive recovery were allowed between the two sets.
  Interventions: Behavioral: exercise training in heart failure with HIIT
- moderate intensity and continuous exercise (Active Comparator): moderate intensity and continuous exercise: 30 minutes at 60% of PPO.
  Interventions: Behavioral: exercise training in heart failure with HIIT

INTERVENTIONS:
Behavioral: exercise training in heart failure with HIIT — to compare MICT vs HIIT 5 days/week during 4 weeks in a Cardiovascular Centre.

SUMMARY:
Purpose: Exaggerated sympathetic nervous system (SNS) activity associated with low heart rate variability (HRV) is considered as a trigger of cardiac arrhythmias and sudden death. Regular exercise training is efficient to improve autonomic balance. In 2013, the investigators published that a single session of an optimized short-high intensity interval exercise with passive recovery (HIIT) protocol was efficient in chronic heart failure (CHF) patients for enhancing vagal tone and to decrease arrhythmias in the 24-h post exercise period when compared to a single session of moderate intensity continuous exercise (MICT). Nevertheless the effects of HIIT training performed on several weeks have never yet been studied on the parameters described by Coumel's triangle (the arrhythmogenic substrate, the trigger factor as premature ventricular contraction and the modulation factors of which the most common is the autonomic nervous system). The aim of this study was to verify the superiority of HIIT to enhance parasympathetic activity, cardiorespiratory fitness and cardiac function when compared to MICT in a short and intense cardiac rehabilitation program.

DETAILED DESCRIPTION:
Before and after the Rehabilitation Program (RP), all patients underwent a 24-hour ECG recording, an echocardiography, a cardiopulmonary exercise test.

The RP consisted of 2 types of exercise training according to the randomization:

1. a short-high intensity interval exercise with passive recovery
2. a classical moderate and continuous exercise training at 60% of peak power output

The RP lasted 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* stable chronic heart failure with NYHA functional class from I to III
* stable left ventricular ejection fraction (LVEF) < 45% over at least 6 months
* stable optimal medical therapy including a beta-blocker and an angiotensin-converting enzyme inhibitor or angiotensin receptor blockers for at least 6 weeks
* ability to perform a maximal cardiopulmonary exercise test
* admitted to the Rehabilitation Centre for a comprehensive Cardiovascular Rehabilitation Program

Exclusion Criteria:

* any relative or absolute contraindications to exercise training according to current recommendations
* fixed-rate pacemaker with heart rate limits set lower than exercise training target
* major cardiovascular event or procedure within the 3 months preceding enrolment
* chronic atrial fibrillation
* heart failure secondary to significant uncorrected primary valve disease (except for mitral regurgitation secondary to left ventricular dysfunction)
* heart failure secondary to congenital heart disease or obstructive cardiomyopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-05-07 (Actual); Primary Completion 2017-10-13 (Actual); Study Completion 2017-10-13 (Actual)

PRIMARY OUTCOMES:
High Frequency power in normalized units (HFnu%) | Change from baseline through study completion, an average of 4 weeks (measured during the night period for stationary signal)
  based on Heart Rate Variability, the power spectral density of the HF (0.15-0.40 Hz, ms2.Hz-1) bands were calculated.

SECONDARY OUTCOMES:
maximal oxygen consumption (VO2peak ml.min.kg) | Change from baseline through study completion, an average of 4 weeks
  VO2 at peak exercise was measured with Cardiopulmonary Exercise Test.
First ventilatory threshold (VT1) (ml.min.kg) | Change from baseline through study completion, an average of 4 weeks
  VO2 at VT1 was measured with Cardiopulmonary Exercise Test.
Heart Rate Recovery (beats per minute, bpm) | Change from baseline through study completion, an average of 4 weeks
  Heart Rate Recovery (with passive recovery) at 1, 2 and 3 minutes after peak exercise (in beats per minute, bpm)
Left Ventricular Ejection Fraction (LVEF, %) | Change from baseline through study completion, an average of 4 weeks
  LV volumes and ejection fraction were calculated from apical recordings by modified biplane Simpson's method.
premature ventricular contraction, (n/24h) | Change from baseline through study completion, an average of 4 weeks
  Ectopic ventricular beats were classified as isolated premature contractions, bigeminy, and salves.
NT-pro-BNP, (ng/L) | Change from baseline through study completion, an average of 4 weeks
  blood sample analysis

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Richard, MD, Principal Investigator — Clinic of Saint-Orens, Cardiovascular and Pulmonary Rehabilitation Center, Saint-Orens-de-Gameville, France; Thibaut Guiraud, PhD, Study Director — Institute of Cardiovascular and Metabolic Diseases, National Institute of Health and Medical Research (INSERM), UMR-1048, Toulouse, France; Florent Besnier, PhD, Study Chair — Clinic of Saint-Orens, Cardiovascular and Pulmonary Rehabilitation Center, Saint-Orens-de-Gameville, France. / Institute of Cardiovascular and Metabolic Diseases, National Institute of Health and Medical Research (INSERM), UMR-1048, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Besnier F, Labrunee M, Richard L, Faggianelli F, Kerros H, Soukarie L, Bousquet M, Garcia JL, Pathak A, Gales C, Guiraud T, Senard JM. Short-term effects of a 3-week interval training program on heart rate variability in chronic heart failure. A randomised controlled trial. Ann Phys Rehabil Med. 2019 Sep;62(5):321-328. doi: 10.1016/j.rehab.2019.06.013. Epub 2019 Jul 25. PMID 31352063

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-03-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT03603743/Prot_SAP_ICF_000.pdf